CLINICAL TRIAL: NCT00662779
Title: Evaluation of the Bronchoprotective Effect of Arformoterol in Children With Exercise Induced Bronchospasm
Brief Title: Bronchoprotective Effect of Arformoterol in Children With Exercise-Induced Bronchospasm (EIB)
Acronym: EIB
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: High number of screen failures-couldn't find qualified subjects in timely manner
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Hengameh Raissy, Pharm.D., Research Associate Professor, Pediatrics, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASRC948; 5-MO1-RR-00997 (Other: GCRC)
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Exercise-induced Bronchospasm
Keywords: asthma; exercise induced bronchospasm; prevention; EIB; children
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 15 mcg arformoterol nebulizer + 1 inhalation of placebo inhalation powder
  Interventions: Drug: arformoterol
- 2 (Active Comparator): 1 inhalation of formoterol fumarate inhalation powder (12 mcg/inhalation) + 2 ml of normal saline nebulizer
  Interventions: Drug: formoterol
- 3 (Placebo Comparator): 1 inhalation of placebo inhalation powder + 2 ml of normal saline nebulizer
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: arformoterol — 15 mcg arformoterol nebulizer
  Other Names: Brand name is Brovana.
  Arms: 1
Drug: formoterol — Formoterol 12 mcg/inhalation, dry powder inhaler
  Other Names: Brand name is Foradil
  Arms: 2
Drug: placebo — placebo dry powder capsules ( lactose) and placebo normal saline for nebulization
  Arms: 3

SUMMARY:
It is our primary hypothesis that pretreatment with arformoterol will provide superior protection against EIB in children with mild-moderate asthma compared to placebo added to the current asthma regimen.

Our secondary hypothesis is that nebulized arformoterol has comparable protection against EIB compared to inhaled formoterol by dry powder inhaler.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, double-dummy, crossover clinical trial which will consist of 5 study visits and will last up to 3 weeks.

Fifteen children 12-17 years of age with asthma and EIB, regardless of current asthma therapy will be eligible for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Children 12-17 years of age
* Physician diagnosed asthma for at least 6 months
* Long term controller medication for at least 4 weeks if any being used
* Females of child-bearing potential agree to use an acceptable form of birth control for the duration of the study
* EIB diagnosed by a positive exercise challenge at screening
* Forced expiratory volume in 1 second (FEV1) greater than 70% of predicted at screening visit

Exclusion Criteria:

* History of cardiac dysfunction
* Inability to perform exercise challenge ( i.e., running on treadmill or performing adequate spirometry)
* Upper respiratory infection in the last 4 weeks
* Severe exacerbation, use of oral steroids, or hospitalization in the last 3 months
* Chronic (greater than 2 weeks) use of a Long Acting Beta Agonist (LABA)
* Pregnancy or lactation
* History of paradoxical bronchospasm with any beta-agonist
* Obesity defined as BMI greater than 30 kg/m2

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
It is our primary hypothesis that pretreatment with arformoterol will provide superior protection against EIB in children with mild-moderate asthma compared to placebo added to the current asthma regimen. | April 2008-April 2010

SECONDARY OUTCOMES:
Our secondary hypothesis is that nebulized arformoterol has comparable protection against EIB compared to inhaled formoterol by dry powder inhaler. | April 2008- April 2010

CONTACTS AND LOCATIONS:
Overall Officials: Hengameh Raissy, Pharm.D., Principal Investigator — University of New Mexico- Pediatric department
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States